CLINICAL TRIAL: NCT02673203
Title: Investigation Into the Effects of Blood Glucose Levels Upon Eating Behavior in Lean and Obese Non-diabetic and Diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1503015469; 1K23DK098286-01A1 (NIH)
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Diabetes
Keywords: glucose monitoring; hunger levels; food intake
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean Healthy Control (Active Comparator): (BMI <25 kg/m2)
  Interventions: Device: Continuous Glucose Monitoring System (CGMS); Behavioral: Food log
- Obese non-diabetic subject (Active Comparator): BMI > 30 kg/m2
  Interventions: Device: Continuous Glucose Monitoring System (CGMS); Behavioral: Food log

INTERVENTIONS:
Device: Continuous Glucose Monitoring System (CGMS) — The CGMS consists of 3 parts: sensor, transmitter and monitor. The small sensor measures the glucose levels from the interstitial tissue. The transmitter is attached on top of the sensor and connects wirelessly to the monitor. The sensor is sterile and comes in an unopened package. It has a plastic wire-like tip that is placed under the skin and continuously measures the glucose levels. One of the study physicians will insert the CGMS wire-like tip under the volunteer's skin with the use of the DEXCOM sensor insertion kit. The transmitter is snapped to the sensor pod and the sensor/transmitter unit will be attached to the skin with an adhesive patch. The monitor is the size of a small hand-held device with a digital screen that displays a graph showing the glucose levels from the previous 4-24 hours.
  Other Names: DEXCOM G4 Platinum
Behavioral: Food log — The Food Record will ask about amount and type of food consumed throughout the day. The participants will also register how hungry they are before the meal and how full they feel after they ate, and type and duration of physical activity

SUMMARY:
To investigate whether the daily glucose profiles as assessed by continuous glucose monitoring for 1 week of normal weight and obese individuals relate to hunger levels and food intake.

DETAILED DESCRIPTION:
To evaluate the effect of blood glucose levels on eating behavior in a population of patients with diabetes in a free-living environment; the investigators plan to study lean healthy control subjects (BMI <25 kg/m2) and obese non-diabetic subjects (BMI > 30 kg/m2).

The participants who qualify will be invited to use the CGMS (DEXCOM G4 Platinum) for up to 7 days. On the visit for placement of the CGMS: 1) the participants will be explained by one of the study physicians how to use a glucometer (FreeStyle or Accu-Check), 2) they will have the CGMS inserted under the skin, and 3) they will be instructed how to fill up the food log (informational brochures are available at the end of the protocol. On the second visit (up to 7 days after the initial visit) the CGMS will be removed from the skin and the glucose meter and food log will be returned to the investigators.

When this study was initially designed, it incorporated 2 additional arms in the study: T1DM and obese T2DM patients. These patients were never recruited for the study.

ELIGIBILITY:
Inclusion Criteria:

* A1c < 10.5 %

Exclusion Criteria:

* BMI <18 (no upper limit),
* Creatinine > 1.5 mg/dL,
* Hgb < 10 mg/dL,
* ALT > 2.5 X ULN,
* untreated thyroid disease,
* uncontrolled hypertension,
* known neurological disorders,
* untreated psychiatric disorders,
* use of antidepressants and psychiatric medications,
* use of weight loss medications in the 6 months prior to the study,
* malignancy,
* smoking,
* current or recent steroid use in last 3 months,
* history of current illicit drug use;
* for women: pregnancy, or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Belfort De Aguiar, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Typical Weight Participants: Participants with a BMI <25 kg/m2.
- Obese Non-diabetic Pariticpants: Non-diabetic participants with a BMI > 30 kg/m2.
Period: Overall Study
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.0) | 40.4 (14.1) | 39 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 11 | 9 | 20
  African American | 1 | 2 | 3
  Hispanic | 2 | 3 | 5
  Asian | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Weight (kg) [Mean (Standard Deviation); unit: kg] | 67.8 (12.0) | 90.6 (12.6) | 79.3 (21.8)
A1c (%) [Mean (Standard Deviation); unit: %] | 5.2 (0.4) | 5.1 (0.7) | 5.1 (0.6)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 23.5 (1.7) | 33.4 (2.2) | 28.3 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Changing Glucose Level
Description: The CGM sensor measures the glucose levels from the interstitial tissue. Presented is the rate of changing glucose level (mg/dl/min).
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl/min
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
mg/dl/min | 0.52 [0.47 to 0.57] | 0.44 [0.38 to 0.49]

2. Primary Outcome: Glucose Peak
Description: The CGM sensor measures the glucose levels from the interstitial tissue. Presented is the glucose peak (mg/dl).
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
mg/dl | 119.5 [111.5 to 127.6] | 121.5 [113.1 to 130.0]

3. Primary Outcome: Glucose Nadir
Description: The CGM sensor measures the glucose levels from the interstitial tissue. Presented is the glucose nadir (mg/dl).
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
mg/dl | 85.1 [79.7 to 90.4] | 87.1 [81.4 to 92.7]

4. Secondary Outcome: Difference in Glucose Peak and Nadir
Description: The CGM sensor measures the glucose levels from the interstitial tissue. Presented is the difference in glucose peak and nadir (mg/dl).
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
mg/dl | 34.3 [29.8 to 38.8] | 33.9 [29.0 to 38.7]

5. Secondary Outcome: Average Daily Hunger Rating
Description: Average daily hunger was measured using a self-report scale. Hunger is measured on a scale from 1-10. 10 is the most hungry, 1 is the least hungry.
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
score on a scale | 5.8 [5.1 to 6.5] | 5.6 [4.9 to 6.4]

6. Secondary Outcome: Nutirion Intake: Energy
Description: Data were collected through food journals. Energy and macronutrient composition were calculated from self-reported food records based on Nutrition Data System for Research (NDS-R). Presented is the average daily energy intake (kcal/day).
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: kcal/day
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
kcal/day | 2251.5 [1841.1 to 2661.8] | 2167.8 [1782.1 to 2553.5]

7. Secondary Outcome: Nutirion Intake: Carbohydrate
Description: Data were collected through food journals. Energy and macronutrient composition were calculated from self-reported food records based on Nutrition Data System for Research (NDS-R). Presented is the average daily carbohydrate intake (g/day).
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: g/day
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
g/day | 261.1 [212.2 to 310.0] | 251.8 [204.5 to 297.1]

8. Secondary Outcome: Nutirion Intake: Fat
Description: Data were collected through food journals. Energy and macronutrient composition were calculated from self-reported food records based on Nutrition Data System for Research (NDS-R). Presented is the average daily fat intake (g/day).
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: g/day
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
g/day | 92.4 [68.3 to 116.5] | 97.5 [74.9 to 120.1]

9. Secondary Outcome: Nutirion Intake: Protein
Description: Data were collected through food journals. Energy and macronutrient composition were calculated from self-reported food records based on Nutrition Data System for Research (NDS-R). Presented is the average daily protein intake (g/day).
Time Frame: 3-5 days
Measure: Least Squares Mean (95% Confidence Interval); unit: g/day
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
Number analyzed (Participants) | 16 | 15
g/day | 99.9 [81.2 to 118.5] | 80.9 [61.9 to 97.9]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for up to 7 days of wearing the CGM.
Arm/Group | Typical Weight Participants | Obese Non-diabetic Pariticpants
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT02673203/Prot_SAP_000.pdf